CLINICAL TRIAL: NCT04940104
Title: Change in Biting Force After Botilinium Toxin Injection and Its Effect on Peri Implant Bone Changes
Brief Title: Change in Biting Force After Botox Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Sara Fikry El Shafei, Principle Investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21-009
Record Dates: First submitted 2021-06-18; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Bruxism
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botox (Experimental)
  Interventions: Drug: Botox Injectable Product
- Control No Botox (No Intervention)

INTERVENTIONS:
Drug: Botox Injectable Product — Botox is a well known neurotoxin that is derived from the bacterium clostridium botulinium. Its therapeutic applications are variable and well documented, alongside its cosmetic applications. There are seven known serotypes of Botox, from A to G, but only two types; A &B, are available for medical and cosmetic uses.
  Arms: Botox

SUMMARY:
Implant rehabilitation is a successful treatment option for edentulous patients. Decreasing bone loss around implants is an important target for all implantologists. It has been shown that pathological forces, such as bruxism, may in fact result in bone loss and eventual implant failure.

Botilinium Toxin is a material of many clinical uses. Beside its cosmetic applications, it has been used in the treatment of masseter muscle hypertrophy.

Purpose: To investigate the effect of botilinium toxin injection on biting forces, and its ultimate effect on peri-implant bone changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a partially edentulous mandible, Kennedy Class I configuration, who are indicated for rehabilitation with partial implant overdenture prostheses, and who complained of Bruxism.

Exclusion Criteria:

* The presence of notable facial asymmetry.
* Severe malocclusion
* Pregnancy
* A history of any serious medical illness
* Drug allergy.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in biting force | 12 months
  Biting force measured using T-Scan

SECONDARY OUTCOMES:
Bone changes around implant | 12 months
  Bone changes using 3D CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in EGYPT, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided